CLINICAL TRIAL: NCT05638750
Title: Twice Weekly Outpatient Rehabilitation Intervention for Young Children With Spinal Muscular Atrophy Treated With Genetic Based Therapies: A Feasibility Study
Brief Title: Outpatient Rehabilitation Intervention for Young Children With SMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Laura McAdam, Medical Director, Child Development Program, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0550
Record Dates: First submitted 2022-11-05; First posted 2022-12-06 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Spinal Muscular Atrophy
Keywords: young children; pediatric; rehabilitation; feasibility study; pilot study
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will participate in the rehabilitation intervention.
  Interventions: Other: Rehabilitation Intervention

INTERVENTIONS:
Other: Rehabilitation Intervention — 12-week treatment intervention & home exercised, then 12-week non-intervention period, follow-up visit at end of non-intervention period.

SUMMARY:
An outpatient rehabilitation program for children (6 months to less than 6 years old) with Spinal Muscular Atrophy (SMA) treated with genetic based therapies is being studied. Participants will participate in a 12-week therapy program where they receive 45 minutes each of occupational therapy and physical therapy each week. Home exercises will also be prescribed to be completed 5 days per week. At the end of the therapy program, there will be a 12-week period of no therapy where only home exercises will be completed. Assessments and program evaluation will occur at the beginning (Week 0) and end of the rehabilitation program (Week 24), then at the end of the no therapy block (week 24).

DETAILED DESCRIPTION:
The standard of care for SMA has historically been physical therapy (PT) and occupational therapy (OT) often focused on strategies that reduce the risk of secondary side effects such as joint tightness. Recently, three genetic based therapies: nusinersen, onasemnogene abeparvovec and risdiplam, have been approved as treatment by Health Canada. Genetic based therapies have provided improvements in physical function for children with SMA. Currently, there is no evidence-based guidance regarding rehabilitation to increase function for children with SMA that have received genetic based therapies. Additionally, there is a lack of published evidence regarding the type of rehabilitation programs and the impact that rehabilitation has on physical function.

An outpatient rehabilitation program for children (6 months to less than 6 years old) with Spinal Muscular Atrophy (SMA) treated with genetic based therapies is being proposed and its feasibility being evaluated. Participants will participate in a 12-week therapy program where they receive 45 minutes each of occupational therapy and physical therapy each week. Home exercises will also be prescribed to be completed 5 days per week. At the end of the therapy program, there will be a 12-week period of no therapy where only home exercises will be completed. Assessments and program evaluation will occur at the beginning (Week 0) and end of the rehabilitation program (Week 24), then at the end of the no therapy block (week 24).

ELIGIBILITY:
Inclusion Criteria:

* SMA (Type I, II or III) diagnosis;
* Receives genetic based therapy;
* Aged 6 months to less than 6 years old;
* Able to participate in weekly therapy at Holland Bloorview (i.e., can attend in-person sessions);
* Able to bring appropriate respiratory equipment to weekly therapy sessions, if required;
* Substitute decision makers (SDMs) must be able to speak and read English;
* Child participant must be able to understand/follow directions in English, as age appropriate;
* SDMs must consent to participate on behalf of their child.

Exclusion Criteria:

* Live outside of Ontario;
* Tracheostomy or use of daytime ventilation (excluding ventilation used during naps).

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Infant Toddler Quality of Life Questionnaire (ITQOL) | Week 0, Week 12, Week 24
  The ITQOL comprises 103 items on 12 scales pertaining to the past four weeks covering physical and psychosocial domains and impact of child health on parents. Scales include: physical functioning, growth and development, bodily pain, temperament/moods, general behaviour, getting along, general health perception, parental-emotional, parental-time, family activities, family cohesion, and change in health. This will be completed for participants ≤3 years old
PedsQL | Week 0, Week 12, Week 24
  he PedsQL parent proxy-report scales measure health-related quality of life in children and adolescents 2-18 years old. PedsQL evaluates quality of life through functioning in physical, emotional, social, and school domains. The parent report for toddlers will be utilized for participants who are 4 years of age and the parent report for young children will be utilized for participants who are 5 years old.
Canadian Occupational Performance Measure (COPM) | Week 0, Week 12, Week 24
  The COPM measures an individual's self-perception of occupational performance on self-care, productivity and leisure. The COPM is used by OTs in initial assessments to set goals and plan treatment focusing on activities that an individual needs, wants or is expected to do. The importance of activities are rated on a 10-point scale (1 = not important at all to 10 = extremely important). The individual selects the five most important activities, which are rated on a 10-point performance scale (1 = not at all able to 10 = able to perform extremely well) and for satisfaction (1 = not at all satisfied to 10 = extremely satisfied). COPM will be completed for all participants.
Goal Attainment Scaling (GAS) | Week 0, Week 12, Week 24
  Goal Attainment Scaling (GAS) is used to evaluate an individual's progress towards client/family goals. Each scale is developed based on assessment and collaboration between the therapist and the client/family. A 5-point scale, ranging from - 2 to +2, is used. A numeric value is assigned to each level of performance. On the original scale, 0 is used to represent the expected level of outcome, with +1 and +2 indicating greater than expected progress and -1 and -2 indicating less than expected progress (reference). Various protocols have been developed to improve the reliability and validity of GAS goals and they can be subjective in nature. GAS will be completed for all participants.
Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND) | Week 0, Week 12, Week 24
  The CHOP-INTEND evaluates the motor skills of patients with SMA Type I aged 3 months to over 4 years. The assessment includes 16 parts. Items are scored on a 4-point scale (0 = no response, 1 = partial level of response, 3 = nearly full level of response, 4= complete level of response). The assessment has good internal consistency (> 0.70) and strong intra-rater reliability (ICC=0.96). CHOP-INTEND will be used for participants who are not independent sitters regardless of age.
Hammersmith Functional Motor Scale - Expanded (HFMSE) | Week 0, Week 12, Week 24
  The 33-item HFMSE assesses the functional motor ability of individuals with SMA who are able to sit and walk using a 3-point scoring system (0 = unable to perform, 1 = performs with modification/adaptation/compensation, 2 = performs without modification/adaptation/compensation). HMFSE will be used for participants who are independent sitters regardless of age.
Bayley Scales of Infant and Toddler DevelopmentTM, 4th Edition | Week 0, Week 12, Week 24
  The Bayley Scale is a developmental assessment tool for diagnosing developmental delays in early childhood (16 days to 42 months) across five domains: cognitive (81 items), language (79 items), motor (103 items), social-emotional (# items) and adaptive behaviour (# items). The entire Bayley Scale can take 30-70 minutes to administer depending on the participant's age. The Bayley will be used with participants ≤3 years old
Peabody Developmental Motor Scales (PDMS), 2nd Edition | Week 0, Week 12, Week 24
  The PDMS is an early childhood motor developmental assessment for gross and fine motor skills. The entire PDMS can take 60-90 minutes to complete. The PDMS will be used with participants >3 years old.
Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), Feasibility of Intervention Measure (FIM) | Week 12
  An implementation outcome measure to evaluate the success of implementation efforts. The AIM, IAM and FIM are each 4-item surveys to evaluate the acceptability, appropriateness and feasibility of the intervention from a personal perspective using a 5-point Likert scale (1 = completely disagree to 5 = completely agree). Internal consistency (α) of the three measures ranged from 0.87 and 0.89, and they take less than five minutes to complete.
Home Exercise Diary | Weeks 1-24
  This purposefully developed form will be completed by the participant's parent/guardian each time the home exercise program is completed. The parent/guardian will be asked to fill out the week of the intervention, day of the week (e.g., Monday), which of the OT/PT exercises were completed (i.e., Yes, No, N/A), and any comments (i.e., about the participant's mood, adverse events, and duration of the exercises). Additionally, the parent/guardian will indicate if any additional activities were completed by the participant in the past week.

OTHER OUTCOMES:
Demographics Survey | Week 0
  This purposefully developed form will capture participant characteristics (e.g., age at intervention commencement (year, month), sex, parent report of genetic condition, genetic based therapies and timing)

CONTACTS AND LOCATIONS:
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ippolito C, Canthiya L, Floreani A, Luckhart K, Hoffman A, McAdam L. Twice-Weekly Outpatient Rehabilitation Intervention for Young Children With Spinal Muscular Atrophy Treated With Genetic-Based Therapies: Protocol for a Feasibility Study. JMIR Res Protoc. 2023 Nov 2;12:e46363. doi: 10.2196/46363. PMID 37917140